CLINICAL TRIAL: NCT00523263
Title: Heparin Bonded and Collagen Coated Polyester or Human Umbilical Vein for Femoropopliteal Bypass: a Prospective Randomised Multicentre Trial.
Brief Title: Dacron vs Dardik for Fem-Pop Bypass
Acronym: DaDa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DaDa-trial
Record Dates: First submitted 2007-08-30; First posted 2007-08-31 (Estimated); Last update posted 2007-08-31 (Estimated); Status verified 2007-08

CONDITIONS: Intermittent Claudication; Arterial Occlusive Diseases; Atheroslerosis
MeSH Terms: conditions — Intermittent Claudication; Arterial Occlusive Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dacron (Active Comparator): Patients receiving polyester above-knee femoro-popliteal bypass
  Interventions: Device: heparin-bonded and collagen coated polyster
- HUV (Active Comparator): patients receiving HUV femoro-popliteal bypass
  Interventions: Device: Human umbilical vein femoro-popliteal bypass

INTERVENTIONS:
Device: heparin-bonded and collagen coated polyster — femoro-popliteal bypass
  Arms: Dacron
Device: Human umbilical vein femoro-popliteal bypass
  Arms: HUV

SUMMARY:
Clinical trial for the comparison of long-term patency of heparin-bonded Dacron and human umbilical vein vascular prostheses in above-knee femoro-popliteal bypass surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 31 to 89
* intermittent claudication
* ABI below 0.8

Exclusion Criteria:

* non elective surgery
* life expectancy below 2 yrs
* contraindication for anticoagulant therapy

Ages: 31 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1996-01; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Primary and primary-assisted bypass patency | 1 - 5 yrs

SECONDARY OUTCOMES:
Secondary bypass patency | 1 - 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: J. Adam van der Vliet, MD, PhD, Principal Investigator — Radboud University Medical Center Nijmegen
Locations (1):
- Radboud UMCN, Dept Vascular Surgery, Nijmegen, Netherlands

REFERENCES:
- [Background] Scharn DM, Oyen WJ, Klemm PL, Verhofstad AA, van der Vliet JA. Thrombogenicity and related biological properties of heparin bonded collagen coated polyester and human umbilical vein prosthetic vascular grafts. J Surg Res. 2006 Aug;134(2):182-9. doi: 10.1016/j.jss.2006.01.025. Epub 2006 Mar 20. PMID 16542682
- [Background] Scharn DM, Oyen WJ, Klemm PL, Wijnen MH, vanderVliet JA. Assessment of prosthetic vascular graft thrombogenicity using the technetium-99m labeled glycoprotein IIb/IIIa receptor antagonist DMP444 in a dog model. Cardiovasc Surg. 2002 Dec;10(6):566-9. doi: 10.1016/s0967-2109(02)00077-7. PMID 12453688
- [Derived] Dirven M, Scharn DM, Blankensteijn JD, van der Vliet JA. Preservation for future use of the autologous saphenous vein during femoro-popliteal bypass surgery is inexpedient. Eur J Vasc Endovasc Surg. 2008 Oct;36(4):420-3. doi: 10.1016/j.ejvs.2008.06.012. PMID 18675557